CLINICAL TRIAL: NCT03155438
Title: Oxidative Stress-related Gene Expression in Cumulus Cells Among Low Responders to Controlled Ovarian Hyperstimulation During in Vitro Fertilization
Brief Title: Oxidative Stress-related Gene Expression in Cumulus Cells Among Low Responders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Porntip Sirayapiwat, Assistant professor, Chulalongkorn University
Other Study IDs: RA60/041; Med Chula IRB No.688/59 (Other: Faculty of Medicine,Chulalongkorn university)
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Low Responder
Keywords: Oxidative stress; Cumulus cell; Controlled ovarian hyperstimulation; In vitro fertilization; Low responder
MeSH Terms: interventions — Transcription, Genetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cumulus cell , Follicular fluid , Blood from IVF patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low responder: Low responder : women aged 25-49 years old with less than 5 oocytes (1-4 oocytes) retrieved during controlled ovarian hyperstimulation
  Oxidative stress-related gene expression and oocyte competence biomarkers will be performed to access the difference between low and normal responders.
  Interventions: Diagnostic Test: Oxidative stress-related gene expression (RNA expression); Diagnostic Test: oocyte competence biomarkers
- Normal responder: Normal responder women aged 25-49 years old with 5-15 oocytes retrieved during controlled ovarian hyperstimulation
  Oxidative stress-related gene expression and oocyte competence biomarkers will be performed to access the difference between low and normal responders.
  Interventions: Diagnostic Test: Oxidative stress-related gene expression (RNA expression); Diagnostic Test: oocyte competence biomarkers

INTERVENTIONS:
Diagnostic Test: Oxidative stress-related gene expression (RNA expression) — Oxidative stress-related gene expression (RNA expression),Superoxide dismutase 1 (SOD1) , SOD2 , Glutathione peroxidase (GPX) and Inducible nitric oxide synthase (iNOS) , measured by Real time PCR technique.
Diagnostic Test: oocyte competence biomarkers — Oocyte competence biomarkers ,GDF9, BMP15, Amphiregulin and CoQ10 measured by ELISA

SUMMARY:
In Vitro Fertilization is considered one of effective treatment for infertile couple. However, some women do not have adequate response to controlled ovarian hyperstimulation, resulting in low response which defined as less than 5 retrieved oocytes. There are studies claiming that live birth rates in these patient lower than normal responder (10-15 retrieved oocytes). Among factors contributing low response, oxidative stress, resulting from increased pro-oxidant and/or reduced antioxidant, is considered to effect the functions of follicles and quality of oocytes. However, there are few studies demonstrating this relation. Objective of our study is to find the difference of oxidative stress-related gene expression in cumulus cell and oocyte competence biomarkers from follicular fluid between low responders and normal responder to controlled ovarian hyperstimulation.

DETAILED DESCRIPTION:
Low response to controlled ovarian hyperstimulation (less than 5 retrieved oocytes) is a problem in some of couple receiving treatment for infertility. Studies showed that success rate in treatment for these patients is lower than normal response group. Among many factors contributing low response, oxidative stress is suspected to be involved in malfunction of follicular environment and oocyte maturation. However, direct relationship between oxidative and oocyte function cannot be studied due to ethical concern, so many studies had studied oocyte's surrounding environment such as cumulus cell and follicular fluid instead.

In our study , we aim to study the difference in level of oxidative stress-related gene expression and oocyte competence biomarkers among low responders and normal responders. For oxidative stress-related gene expression of cumulus cell , we will measure mRNA expression by quantitative PCR for Superoxide dismutase 1 (SOD1) , SOD2 , Glutathione peroxidase (GPX) and Inducible nitric oxide synthase (iNOS) . For oocyte competent biomarkers, we will use ELISA technique to measure the level of GDF(, BMP15, Amphiregulin and CoQ10 in follicular fluid.

Sample size calculation was done with data from study performed by Donnabela et al , which found that Mean SOD gene expression in control group was 2.06 2-Δ ΔCT (SD = 0.53) . The formula for comparing two different mean was used with expectation that low responders group would have lower SOD gene expression by 20%.:

n/group = 2(Z α/2 + Z β)2 σ2 / (X̅ 1- X̅ 2)2

α = 0.05 , β = 0.2 Z α/2 = Z0.05/2 = 1.96 (two tail) Z β = Z0.8 = 0.84

Mean in group1 (X̅ 1) = 2.06, SD. in group1 (σ₁) = 0.53 Mean in group2 (X̅ 2) = 1.64, SD. in group2 (σ₂)= 0.53 Sample size: Group1 (n₁) = 25, Group2 (n₂) = 25 Total number is 56 patients (added 10% for possible data loss)

Statistical analysis

1. Mean and Standard deviation will be used for descriptive data.
2. Mann-Whitney U test , unpaired t-test and chi square will be used as appropriate
3. p value less than 0.05 is considered statistical significant.

ELIGIBILITY:
Inclusion Criteria:

* Low responder : women aged 25-49 years old with less than 5 oocytes (1-4 oocytes) retrieved during controlled ovarian hyperstimulation
* Normal responder women aged 25-49 years old with 5-15 oocytes retrieved during controlled ovarian hyperstimulation

Exclusion Criteria:

* Active ovarian pathology ( ovarian cyst or tumor)
* Basal FSH more than 20 IU/L or Antimullerian hormone less than 0.5 ng/ml
* Ovarian hyperstimulation syndrome

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women aged 25-49 years old , who receiving care at infertile clinic ,King Chulalongkorn Memorial hospital
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress-related gene expression | June 2017-May 2018
  mRNA expression by quantitative PCR for Superoxide dismutase 1 (SOD1) SOD2 , Glutathione peroxidase (GPX) and Inducible nitric oxide synthase (iNOS).

SECONDARY OUTCOMES:
oocyte competent biomarkers | June 2017-May 2018
  ELISA technique to measure the level of GDF9, BMP15, Amphiregulin and CoQ10 in follicular fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Porntip Sirayapiwat, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine ,Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polyzos NP, Sunkara SK. Sub-optimal responders following controlled ovarian stimulation: an overlooked group? Hum Reprod. 2015 Sep;30(9):2005-8. doi: 10.1093/humrep/dev149. Epub 2015 Jul 21. PMID 26202582
- [Background] Oudendijk JF, Yarde F, Eijkemans MJ, Broekmans FJ, Broer SL. The poor responder in IVF: is the prognosis always poor?: a systematic review. Hum Reprod Update. 2012 Jan-Feb;18(1):1-11. doi: 10.1093/humupd/dmr037. Epub 2011 Oct 10. PMID 21987525
- [Background] Agarwal A, Aponte-Mellado A, Premkumar BJ, Shaman A, Gupta S. The effects of oxidative stress on female reproduction: a review. Reprod Biol Endocrinol. 2012 Jun 29;10:49. doi: 10.1186/1477-7827-10-49. PMID 22748101
- [Background] Nunez-Calonge R, Cortes S, Gutierrez Gonzalez LM, Kireev R, Vara E, Ortega L, Caballero P, Rancan L, Tresguerres J. Oxidative stress in follicular fluid of young women with low response compared with fertile oocyte donors. Reprod Biomed Online. 2016 Apr;32(4):446-56. doi: 10.1016/j.rbmo.2015.12.010. Epub 2016 Jan 14. PMID 26805046
- [Background] Dumesic DA, Meldrum DR, Katz-Jaffe MG, Krisher RL, Schoolcraft WB. Oocyte environment: follicular fluid and cumulus cells are critical for oocyte health. Fertil Steril. 2015 Feb;103(2):303-16. doi: 10.1016/j.fertnstert.2014.11.015. Epub 2014 Dec 10. PMID 25497448
- [Background] Wu YT, Tang L, Cai J, Lu XE, Xu J, Zhu XM, Luo Q, Huang HF. High bone morphogenetic protein-15 level in follicular fluid is associated with high quality oocyte and subsequent embryonic development. Hum Reprod. 2007 Jun;22(6):1526-31. doi: 10.1093/humrep/dem029. Epub 2007 Mar 8. PMID 17347167
- [Background] Gode F, Gulekli B, Dogan E, Korhan P, Dogan S, Bige O, Cimrin D, Atabey N. Influence of follicular fluid GDF9 and BMP15 on embryo quality. Fertil Steril. 2011 Jun;95(7):2274-8. doi: 10.1016/j.fertnstert.2011.03.045. Epub 2011 Apr 15. PMID 21496799
- [Background] Liu N, Ma Y, Li R, Jin H, Li M, Huang X, Feng HL, Qiao J. Comparison of follicular fluid amphiregulin and EGF concentrations in patients undergoing IVF with different stimulation protocols. Endocrine. 2012 Dec;42(3):708-16. doi: 10.1007/s12020-012-9706-z. Epub 2012 Jun 8. PMID 22678853
- [Background] Bergandi L, Basso G, Evangelista F, Canosa S, Dalmasso P, Aldieri E, Revelli A, Benedetto C, Ghigo D. Inducible nitric oxide synthase and heme oxygenase 1 are expressed in human cumulus cells and may be used as biomarkers of oocyte competence. Reprod Sci. 2014 Nov;21(11):1370-7. doi: 10.1177/1933719114525268. Epub 2014 Mar 7. PMID 24607880
- [Result] Donabela FC, Meola J, Padovan CC, de Paz CC, Navarro PA. Higher SOD1 Gene Expression in Cumulus Cells From Infertile Women With Moderate and Severe Endometriosis. Reprod Sci. 2015 Nov;22(11):1452-60. doi: 10.1177/1933719115585146. Epub 2015 May 6. PMID 25947891